CLINICAL TRIAL: NCT01120392
Title: Virtual Reality in Motor Performance and Quality of Life in Patients With Parkinson's Disease
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Federal University of Bahia (Other)
Responsible Party: Principal Investigator, Ailton de Souza Melo, PhD, Federal University of Bahia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DNEP
Record Dates: First submitted 2010-05-10; First posted 2010-05-11 (Estimated); Last update posted 2011-12-07 (Estimated); Status verified 2011-12

CONDITIONS: Parkinson Disease
Keywords: Parkinson's disease; Physical therapy; Virtual Reality; Quality of life; Motor performance
MeSH Terms: conditions — Parkinson Disease | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment group - Nintendo wii. (Experimental)
  Interventions: Other: treatment with Nintendo wii.
- conventional - Physical Therapy (Active Comparator)
  Interventions: Other: Physical therapy conventional.

INTERVENTIONS:
Other: treatment with Nintendo wii. — Participants Will receive treatment with Nintendo Wii over one months. These Patients Will Be subjected to mobilization of stem and stretching. Then Will Be Submitted to Nintendo wii games. Will Be Submitted This group three times a week to a treatment protocol with boxing exercises with wii sports and wii fit
  Arms: Treatment group - Nintendo wii.
Other: Physical therapy conventional. — Conventional exercises used with the same goals for the group with wii
  Arms: conventional - Physical Therapy

SUMMARY:
Treatment with Nintendo wii is higher to physical therapy conventional in the quality of life and motor performance in patients with Parkinson's disease.

DETAILED DESCRIPTION:
The aim of this study is to assess if the treatment of rehabilitation with Nintendo wii is higher to the conventional in the quality of life and motor performance in patients with Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Parkinson's disease
* Both the sex with age between 50 and 80 years
* To be in it I serve as apprentice of 1 the 3,0 in the scale of Hoehn Yahr

Exclusion Criteria:

* Cognitive impairment
* Poorly controlled arterial hypertension
* Poorly controlled Cardiopathy

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-05; Primary Completion 2011-09 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Quality of life | 4 weeks (Baseline and after four weeks)
  Parkinson's disease questionnaire (PDQ-39)
Motor performance | 4 weeks (Baseline and after four weeks)
  the Unified Parkinson's Disease Rating Scale (UPDRS.)

CONTACTS AND LOCATIONS:
Overall Officials: Ailton Melo, PhD, Principal Investigator — UFBA- DINEP
Locations (1):
- Ambulatorio Magalhães Neto, Salvador, Estado de Bahia, Brazil

REFERENCES:
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886